CLINICAL TRIAL: NCT01483729
Title: A Relative Bioavailability Study of Danoprevir and Ritonavir in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NP27945; RPU425UD-114254 (Other: PRA International)
Record Dates: First submitted 2011-11-30; First posted 2011-12-01 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — danoprevir; Ritonavir

ARMS (6):
- Part 1 A (Active Comparator)
  Interventions: Drug: danoprevir; Drug: ritonavir
- Part 1 B (Experimental)
  Interventions: Drug: danoprevir; Drug: ritonavir
- Part 1 C (Experimental)
  Interventions: Drug: danoprevir; Drug: ritonavir
- Part 2 D (Active Comparator)
  Interventions: Drug: danoprevir; Drug: ritonavir
- Part 2 E (Experimental)
  Interventions: Drug: danoprevir; Drug: ritonavir
- Part 2 F (Experimental)
  Interventions: Drug: danoprevir; Drug: ritonavir

INTERVENTIONS:
Drug: danoprevir — Phase 3 Tablet Formulation 1, single oral dose
  Arms: Part 1 B
Drug: danoprevir — Phase 3 Tablet Formulation 2, single oral dose
  Arms: Part 1 C
Drug: danoprevir — Reference Phase 2 Tablet Formulation, single oral dose
  Arms: Part 1 A; Part 2 D; Part 2 E; Part 2 F
Drug: ritonavir — Test Formulation 1, single oral dose
  Arms: Part 2 E
Drug: ritonavir — Test Formulation 2, single oral dose
  Arms: Part 2 F
Drug: ritonavir — Reference Formulation, single oral dose
  Arms: Part 1 A; Part 1 B; Part 1 C; Part 2 D

SUMMARY:
This single dose, randomized, open-label, 6 sequence, 3-period, crossover study will evaluate the relative bioavailability of danoprevir and ritonavir in healthy volunteers. In Part 1, subjects will be randomized to receive single oral doses of one of three tablet formulations of danoprevir plus the reference ritonavir formulation, with an at least 7-day washout between periods. In Part 2, subjects will be randomized to receive single oral doses of one of three tablet formulations of ritonavir plus the reference formulation of danoprevir, with at least a 7-day washout betwen periods. The anticipated time on study is up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, 18 to 45 years of age inclusive
* Body mass index 18.0 - 32.0 kg/m2, weight >/= 50 kg
* Healthy status will be defined as absence of evidence of any active or chronic disease following a detailed medical and surgical history and a complete physical examination
* Non-smoker
* Medical history without major, recent or ongoing pathology
* Females of childbearing potential and males and their female partners of childbearing potential must agree to use 2 forms of contraception (barrier form plus intrauterine device and spemicide) during the study and for 90 days after the last drug administration

Exclusion Criteria:

* Pregnant or lactating women or males with female partners who are pregnant or lactating
* Positive results for drugs of abuse at screening or prior to admission to the clinical site during any study period
* Positive for hepatitis B, hepatitis C or HIV infection
* Use of hormonal contraceptives (birth control pills, injectable, implantable devices) within 30 days before the first dose of study medication
* Routine use of more than 2 g of acetaminophen daily
* History of clinically significant drug allergy (such as anaphylaxis) or hepatotoxicity
* History of hypersensitivity to danoptevir, ritonavir, or other protease inhibitors
* History (within 3 months of screening) of alcohol consumption exceeding 2 standard drinks per day on average
* Current enrollment or participation in a clinical trial of an experimental medication or medical device within 3 months of screening unless agreed upon by the Sponsor

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Part 1: Danoprevir bioavailabilty (Tablet Formulation 1) in combination with ritonavir (reference formulation): Area under the concentration-time curve (AUC) | 24 hours
Part 1: Danoprevir bioavailability (Tablet Formulation 2) in combination with ritonavir (reference formulation): Area under the concentration-time curve (AUC) | 24 hours
Part 2: Ritonavir bioavailability (Test Formulation 1) in combination with danoprevir (refernce formulation): Area under the concentration-time curve (AUC) | 24 hours
Part 2: Ritonavir bioavailability (Test Formulation 2) in combination with danoprevir (reference formulation): Area under the concentration-time curve (AUC) | 24 hours

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Christchurch, New Zealand